CLINICAL TRIAL: NCT02395575
Title: Prospective Study Evaluating the Clinical Impact of the Breast Cancer Intrinsic Subtype-Prosigna Test (Assay) in the Management of Early-stage Breast Cancers
Brief Title: A Study of Clinical Outcomes for the NanoString® Technologies Prosigna™ Gene Signature Assay
Status: Completed | Type: Observational
Sponsor: NanoString Technologies, Inc. (Industry)
Collaborators: Institut Curie (Other)
Responsible Party: Sponsor
Other Study IDs: PTL-10018
Record Dates: First submitted 2015-03-17; First posted 2015-03-23 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — FFPE breast tumor tissue samples
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective of this study is to evaluate the impact of the result of the Prosigna Test (assay) on the therapeutic decision of adjuvant therapy (chemotherapy and hormone therapy) in patients suffering from early-stage breast cancer.

DETAILED DESCRIPTION:
The secondary objectives will consist of:

* The evaluation of the confidence in the therapeutic indications of the practitioners before and after the test (assay) results, and by subgroups of cancers
* The evaluation of the rate of secondary effects of chemotherapy,
* The evaluation of the emotional state of patients faced with the therapeutic decision, of their degree of anxiety and of their functional status before and after the Prosigna test (assay) results

ELIGIBILITY:
Inclusion Criteria:

* Resected node-negative, estrogen-receptor-positive, HER2-negative early- stage invasive breast cancer (T1-T2, N0, pN0 (i+), pN0 (mol+), M0)

  * Estrogen receptor status will be evaluated by Immunohistochemistry (IHC) and more than 1% of stained tumor cells will be considered positive.
  * HER2 status will be evaluated by IHC (0 or 1+, or 2+ will be considered negative) and by in-situ fluorescence hybridization.
* Postmenopausal women defined as:

  * Natural Amenorrhea > 12 months, regardless of age
  * Bilateral oophorectomy, regardless of age (the oophorectomy must have been carried out at least 4 weeks before entering the study)
  * Radiological castration with amenorrhea > 3 months, regardless of age
  * Hysterectomy and postmenopausal blood levels
* Able to give consent
* Eligible for treatment of breast cancer with adjuvant chemotherapy
* ECOG performance status of 0 or 1

Exclusion Criteria:

* Tumor size T3-T4
* Non-invasive breast cancer (e.g., Paget's disease, DCIS)
* Tumors with nodes that are not N0, pN0 (i+), or pN0 (mol+)
* Tumors that are estrogen-receptor negative or HER2 positive
* Have metastatic disease
* Unable to give informed consent
* Unable to complete patient reported outcome surveys
* Have contraindications for adjuvant chemotherapy

  * Age, performance status, significant comorbidities
* ECOG performance status > 1

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Postmenopausal women with node-negative, estrogen-receptor positive, HER2-negative early-stage breast cancer. Investigators will offer enrollment to consecutively seen women who meet the entry criteria,
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2015-03; Primary Completion 2016-12 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
The proportion of patients whose choice of treatment is changed as a result of receiving the Prosigna test results. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Roman Rouzier, MD, PhD, Principal Investigator — Institut Curie
Locations (1):
- Institut Curie, Paris, France

IPD SHARING:
Plan to Share IPD: No